CLINICAL TRIAL: NCT01501019
Title: Effects of Exercise Training in Primary Sjogren´s Syndrome, Myositis and Takayasu's Arteritis
Brief Title: Exercise in Sjogren, Myositis and Takayasu's Arteritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exercise in Autoimmunity
Record Dates: First submitted 2011-11-29; First posted 2011-12-29 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Primary Sjogren´s Syndrome; Myositis
MeSH Terms: conditions — Myositis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sjogren and Myositis Control (no control for takayasu's) (No Intervention)
- Sjogren, Myositis and Takayasu's Trained (Experimental)
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — "Sjöegren arm": 30-60 minutes of combined aerobic and strength exercises, twice a week, moderate intensity.
  "Myositis arm": 30 minutes of resistance training combined partial blood flow restriction, twice a week, low intensity.
  "Takayasu's arteritis arm": 30-50 minutes of aerobic, twice a week, moderate intensity.
  Arms: Sjogren, Myositis and Takayasu's Trained

SUMMARY:
Exercise may improve physical capacity and health parameters in Primary Syndrome´s Sjogren, Myositis and Takayasu's Arteritis.

Therefore, this study aims to investigate the role of an exercise training program in patients with Primary Syndrome´s Sjogren, Myositis and Takayasu's Arteritis.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive
* Stable drugs regime for at least three months

Exclusion Criteria:

* Other rheumatic diseases
* Physical disability that prevent the patient to perform the physical tests
* Severe pulmonary disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Aerobic Capacity | Twelve weeks
  Maximum Oxygen Consumption (VO2Max)
Muscle strength | Twelve weeks
Quality of life | Twelve weeks

SECONDARY OUTCOMES:
Serum anti-inflammatory cytokines | Twelve weeks
  Interleukin-10
Serum pro-inflammatory cytokines | Twelve weeks
  Interleukin-1 (IL-1), interleukin-6 (IL-6), tumor necrosis factor-a (TNF-a)
Serum inflammatory markers | Twelve weeks
  erythrocyte sedimentation rate (ESR), c-reactive protein (CRP), aldolase

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo School of Medicine Clinical Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Mattar MA, Gualano B, Perandini LA, Shinjo SK, Lima FR, Sa-Pinto AL, Roschel H. Safety and possible effects of low-intensity resistance training associated with partial blood flow restriction in polymyositis and dermatomyositis. Arthritis Res Ther. 2014 Oct 25;16(5):473. doi: 10.1186/s13075-014-0473-5. PMID 25344395